CLINICAL TRIAL: NCT00079950
Title: Efficacy and Safety Evaluation of Pegamotecan (PEG-camptothecin) in Advanced or Metastatic Soft Tissue Sarcoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Senior Director, Regulatory Affairs, Enzon Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-9009
Record Dates: First submitted 2004-03-18; First posted 2004-03-22 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Sarcoma, Soft Tissue
Keywords: soft; sarcoma; metastatic
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — pegamotecan

INTERVENTIONS:
Drug: Pegamotecan

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Pegamotecan (Peg-Camptothecin) in patients with Advanced or Metastatic Soft Tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of soft tissue sarcoma with measurable disease.
* Target tumors outside prior radiation field(s).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate hematologic profile, as determined by hemoglobin, platelet, and neutrophil count.
* Adequate renal function
* Adequate liver function
* No history of hemorrhagic cystitis or evidence of microscopic hematuria
* Capable of understanding the protocol requirements and risks and providing written informed consent.
* Either 0 or 1 prior chemotherapy regimens

Exclusion Criteria:

* Subject has a diagnosis of gastrointestinal stromal tumors.
* Concurrent serious medical illness unrelated to tumor within the past 6 months.
* Known chronic infectious disease, such as AIDS or hepatitis.
* Positive screening pregnancy test or is breast-feeding.
* A female or male subject of reproductive capacity unwilling to use methods appropriate to prevent pregnancy during the course of this study.
* Receiving concurrent chemotherapy, radiotherapy, or surgery, or has received wide field radiation within the previous 4 weeks.
* History of another active malignancy (except non-melanoma skin cancer and carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for the last 2 years.
* Known or clinically suspected brain metastases.
* Received more than one prior treatment regimen (excluding adjuvant or neoadjuvant therapy) for soft tissue sarcoma.
* Received any investigational drug within the last 30 days.
* Not fully recovered from any prior surgery (at least 4 weeks recovery period for major surgery), and from any reversible side effects related to the administration of cytotoxic chemotherapy or radiation therapy.
* Received a prior camptothecin analog (e.g., topotecan, irinotecan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Century City Hospital, Los Angeles, California
  - Pennsylvania Oncology Hematology Association, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Institute for Drug Development Cancer Therapy and Research Center, San Antonio, Texas